CLINICAL TRIAL: NCT00598689
Title: Efficacy, Tolerability and Comfort of GenTeal and GenTeal Gel, (0.3% Hypromellose) in the Pre- and Post- Operative Treatment of Patients Undergoing LASIK Surgery
Brief Title: GenTeal in Perioperative Treatment of Laser Assisted in Situ Keratomileusis LASIK Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, David Bogorad, Professor and Vice Chairman, Director, Refractive Surgery Service, Department of Ophthalmology, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-09-052
Record Dates: First submitted 2008-01-10; First posted 2008-01-22 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Corneal Epithelium Defect
Keywords: LASIK; Ocular Lubricants; Corneal Epithelium; Wound Healing
MeSH Terms: interventions — Hypromellose Derivatives

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lubricant (Experimental): Patients scheduled to receive LASIK surgery and randomized to receive 0.3% hypromellose ophthalmic solution prior to surgery.
  Interventions: Drug: 0.3% hypromellose
- No Lubricant (No Intervention): Patients scheduled to receive LASIK surgery and randomized to receive no intervention of 0.3% hypromellose ophthalmic solution prior to surgery

INTERVENTIONS:
Drug: 0.3% hypromellose — 0.3% hypromellose four times a day for 5 days prior to LASIK surgery
  Other Names: Genteal Gel
  Arms: Lubricant

SUMMARY:
GenTeal gel is an artificial tear gel used to lubricate the surface of the eye. This study will evaluate the effect of GenTeal gel on comfort following LASIK surgery. Participants will be asked to come to the clinic for three regularly scheduled visits after LASIK surgery: Day 1 (one day after LASIK surgery), Day 7 (one week follow-up), and Day 30 (one month follow-up). Participants will be asked to complete a questionnaire regarding eye comfort during each follow up visit. Participants will be randomly assigned to one of two groups, one of which will receive Genteal Gel four times a day for five days prior to surgery. The other group will receive no preoperative gel or lubricant, which has been our standard approach for many years.

DETAILED DESCRIPTION:
LASIK (Laser Keratomileusis in Situ) is a frequently performed procedure to reduce the refractive error of the eye so as to minimize the subsequent need for eyeglasses or contact lenses. The procedure requires the creation of a superficial corneal flap, usually with an instrument known as a microkeratome. During the creation of the flap with a microkeratome, the corneal epithelium is typically subjected to sliding stresses which occasionally cause disruption of the epithelial surface, a complication with potentially serious adverse effect on the post operative visual acuity. As well, shortly before the creation of the flap, the patient is often dilated and invariably treated with topical anesthetics. These agents, and their preservatives, can have a negative effect on corneal epithelial integrity, right before the epithelium must withstand the passage of the microkeratome. Therefore, it is imperative that the epithelium be in the best possible condition prior to the LASIK procedure. For this reason, ocular lubricants may be used for a period of time prior to surgery in order to maximize epithelial health.

In the immediate post-operative period the bond between the newly created flap and the underlying corneal stroma is weak, and the epithelium has just been subjected to the pharmacologic and mechanical stresses noted above. It is imperative that the surface continuity of the epithelium between the edge of the flap and the surrounding surface be restored as rapidly as possible, as reestablishment of an intact epithelial surface minimizes the risks of flap shift, epithelial ingrowth, and infection. For all these reasons, it is a generally accepted standard of care to use aggressive ocular lubrication during the post-operative period in order to maximize the speed of epithelial recovery.

GenTeal Lubricant Eye Drops and GenTeal Gel, (0.3% hypromellose, Novartis Ophthalmics, Basel, Switzerland) provide a natural alternative to preservative-free treatments, with a sodium perborate preservative system and long-lasting action due to the carbomer gelling agent. The perborate preservative, which breaks down to water and oxygen on the ocular surface, essentially delivers a preservative-free lubricant to the eye. This makes the GenTeal products attractive agents for use in the LASIK perioperative period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 60
2. Both sexes
3. Any race
4. Seeking LASIK surgery at the Medical College of Georgia (MCG)/Eye Care One
5. Meeting all established criteria for appropriateness for LASIK established by MCG/Eye Care One

Exclusion Criteria:

1. Any corneal pathology including scars, prior herpes keratitis, prior corneal transplant
2. Any immunocompromised state including diabetes mellitus, cancer, HIV infection, or Hepatitis B or C.
3. Failure to meet all established criteria for appropriateness for LASIK established by MCG/Eye Care One

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David D Bogorad, M.D, Principal Investigator — Augusta University
Locations (1):
- EyeCare One, Augusta, Georgia, United States

REFERENCES:
- [Background] Samuel MA, Kaufman SC, Ahee JA, Wee C, Bogorad D. Diffuse lamellar keratitis associated with carboxymethylcellulose sodium 1% after laser in situ keratomileusis. J Cataract Refract Surg. 2002 Aug;28(8):1409-11. doi: 10.1016/s0886-3350(02)01266-x. PMID 12160811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 subjects were recruited over a period of four months. Subjects were recruited from the pool of patient scheduled to have Laser Assisted in situ Keratomileusis (LASIK) surgery at the Medical College of Georgia/Eye Care One Laser Vision Center, Augusta, Georgia.
Pre-assignment Details: Subjects were stratified based on smoking status.
Period: Overall Study
Arm/Group | Lubricant | No Lubricant
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Consented subjects with a best corrected visual acuity of 20/40 or better in each eye.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubricant | No Lubricant | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 14 | 13 | 27
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Number of subjects with best corrected visual acuity of 20/40 or better in each eye [Number; unit: participants] | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Epithelial Healing After Laser Assisted in Situ Keratomileusis (LASIK) Surgery
Description: Assess whether preoperative GenTeal Gel enhances epithelial healing after LASIK surgery within the first post-operative week, compared to control (no preoperative lubricant). Healing of the area of the cornea covering the radius of the sectioned into clock hours 0 - 12 where 0 hours equals no healing and 12 hours equals complete healing.
Time Frame: Day 1, End of Week 1
Population: Subjects that completed LASIK surgery.
Measure: Mean (Standard Deviation); unit: Clock Hours
Arm/Group | Lubricant | No Lubricant
Number analyzed (Participants) | 40 | 40
Clock Hours
  Day 1 post LASIK surgery | 4.3 (3.8) | 3.5 (3.0)
  Week 1 post LASIK surgery | 9.2 (1.5) | 9.0 (1.8)

2. Secondary Outcome: Post Operative Pain Level
Description: Assess whether preoperative GenTeal Gel alleviates post operative pain in LASIK surgery patients compared to control (no preoperative lubricant) as measured by patient completion of the Universal Pain Assessment Tool (moderate), a ten point scale with 0 being no pain and 10 being the worst pain possible. Data on the level of pain only in the right eye will be collected.
Time Frame: Day 1, End of Week 1
Population: Subjects that completed LASIK surgery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubricant | No Lubricant
Number analyzed (Participants) | 40 | 40
units on a scale
  Day 1 post LASIK Surgery | 5.2 (2.6) | 5.4 (2.5)
  End of Week 1 post LASIK surgery | 2.8 (2.1) | 3.1 (2.6)

3. Secondary Outcome: Tolerability and Alleviation of Post-operative Pain in LASIK Surgery
Description: A comparison of subjective comfort level defined as tolerability and alleviation of post-operative pain experienced as a result of post-operative application of GenTeal drops. Subjective pain level was measured on a 10 point likert scale where 0 = no pain and 10 = worst pain possible. A lower score at Week 1 as compared to Day 1 was considered improved. A same score or higher at week 1 as compared to day 1 was considered no improvement.
Time Frame: Week 1 post surgery
Population: Subjects randomized to either group and completed LASIK surgery.
Measure: Number; unit: percentage of subjects
Arm/Group | Lubricant | No Lubricant
Number analyzed (Participants) | 40 | 40
percentage of subjects
  Comfort level iimproved at Week 1 | 80 | 87.5
  Comfort level not improved at week 1 | 20 | 12.5

ADVERSE EVENTS:
Arm/Group | Lubricant | No Lubricant
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No